CLINICAL TRIAL: NCT01158560
Title: McFlu2 COLD3 Prevention: A Randomized, Placebo-controlled, Double Blind Trial of Vitamin D and Health Advice for the Prevention of Upper Respiratory Tract Infections in McMaster University Students
Brief Title: A Trial of Vitamin D and Health Advice for the Prevention of Upper Respiratory Tract Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: McFlu2 10-313
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Upper Respiratory Tract Infections; Rhinovirus; Infections
Keywords: upper respiratory tract infections; rhinovirus infections; vitamin D
MeSH Terms: conditions — Respiratory Tract Infections; Infections | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D and gargling (Experimental): Participants will be given a weekly dose of 10,000 IU of vitamin D3 (oral capsule) and asked to gargle with tap water twice daily
  Interventions: Dietary Supplement: cholecalciferol (vitamin D3); Behavioral: Gargling
- Vitamin D and general health advice (Experimental): Participants will be given a weekly dose of 10,000 IU of vitamin D3 (oral capsule) and will receive general health advice in place of gargling advice
  Interventions: Dietary Supplement: cholecalciferol (vitamin D3)
- Placebo and general health advice (Placebo Comparator): Participants will be given an aesthetically matched placebo capsule to take once weekly and will be given general health advice in place of gargling advice.
  Interventions: Dietary Supplement: Placebo
- Placebo and gargling (Placebo Comparator): Participants will be given an aesthetically matched placebo capsule to take once weekly and will be asked to gargle with tap water twice daily
  Interventions: Behavioral: Gargling; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: cholecalciferol (vitamin D3) — oral capsule, 10,000 IU/week vitamin D3 for 6-8 weeks
  Arms: Vitamin D and gargling; Vitamin D and general health advice
Behavioral: Gargling — gargling with tap water, twice daily
  Arms: Placebo and gargling; Vitamin D and gargling
Dietary Supplement: Placebo — matched placebo for active vitamin D
  Arms: Placebo and gargling; Placebo and general health advice

SUMMARY:
The specific objectives of this investigation are to assess the effectiveness of daily gargling and vitamin D supplementation as preventative measures against incident upper respiratory tract infection (URTI) in students attending McMaster University. Investigators hypothesize that

1. Vitamin D3 supplementation will decrease the incidence of symptomatic upper respiratory tract infections in university students
2. Gargling will decrease the incidence of symptomatic upper respiratory tract infections in university students.

DETAILED DESCRIPTION:
In the current study, we propose investigating the roles of vitamin D supplementation and of regular gargling to prevent URTI/ILI. Vitamin D may be an important factor in respiratory health. Observational studies have associated low serum 25(OH)D levels with more frequent and more severe respiratory infections. However, evidence is lacking that replacement of vitamin D decreases respiratory infections. Four interventional studies of vitamin D supplementation have noted a reduction in respiratory infections, with an estimated 5-25% reduction, but results were not statistically significant.

In Japanese populations, gargling has been found to significantly reduce the incidence of upper respiratory tract infections by approximately 35% (Satomura et al., 2005). This intervention has not been studied in different populations but may be a useful personal practice to reduce URTI.

We propose a 2X2 factorial, randomized, placebo-controlled trial of vitamin D/placebo and gargling/no gargling to study the effects of vitamin D supplementation and gargling on upper respiratory tract infections in McMaster students. This study will be conducted over two years, during September and October of each study year, to capture the natural peak in rhinovirus activity.

ELIGIBILITY:
Inclusion Criteria:

* Current or part-time student at McMaster University
* 17 year of age or older
* Currently living:

  i. In residence or, ii. Off-campus with at least one student housemate
* Willing and able to sign an informed consent

Exclusion Criteria:

* Students who do not meet the inclusion criteria
* Currently living at home with parents
* History or diagnosis of hypercalcemia
* Diagnosis of parathyroid disorder (hyper or hypo)
* Diagnosis of chronic kidney disease
* Use of anticonvulsants
* Malabsorption syndromes
* Diagnosis of sarcoidosis
* Currently pregnant or planning a pregnancy
* Inability to swallow capsules

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The number of individuals with self-reported URTI in each of the intervention and control groups | Over the course of 8 weeks spanning September and October

SECONDARY OUTCOMES:
The severity of symptoms in each of the intervention and control groups | Symptoms will be monitored daily for 7 days and a follow-up survey will be administered at day 14
  Daily symptom surveys will be completed for 7 consecutive days follwing the onset of illness. A follow-up survey will be administered at day 14. Surveys will score the severity of symptoms.
Duration of symptoms in each of the intervention and control groups | Symptoms will be monitored daily for 7 days and a follow-up survey will be administered at day 14
  Daily symptom surveys will be completed for 7 consecutive days follwing the onset of illness. A follow-up survey will be administered at day 14.

CONTACTS AND LOCATIONS:
Overall Officials: Marek Smieja, MD, MSc, PhD, FRCPC, Principal Investigator — St. Joseph's Healthcare, McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Jefferson T, Dooley L, Ferroni E, Al-Ansary LA, van Driel ML, Bawazeer GA, Jones MA, Hoffmann TC, Clark J, Beller EM, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2023 Jan 30;1(1):CD006207. doi: 10.1002/14651858.CD006207.pub6. PMID 36715243
- [Derived] Jefferson T, Del Mar CB, Dooley L, Ferroni E, Al-Ansary LA, Bawazeer GA, van Driel ML, Jones MA, Thorning S, Beller EM, Clark J, Hoffmann TC, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2020 Nov 20;11(11):CD006207. doi: 10.1002/14651858.CD006207.pub5. PMID 33215698
- [Derived] Goodall EC, Granados AC, Luinstra K, Pullenayegum E, Coleman BL, Loeb M, Smieja M. Vitamin D3 and gargling for the prevention of upper respiratory tract infections: a randomized controlled trial. BMC Infect Dis. 2014 May 19;14:273. doi: 10.1186/1471-2334-14-273. PMID 24885201